CLINICAL TRIAL: NCT04299308
Title: Acute Exercise Response On Brain Imaging and Cognition
Brief Title: Acute Exercise and the Cerebral Metabolic Response in Aging and Alzheimer's Disease
Acronym: AEROBIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00142140; 1R01AG062548-01A1 (NIH)
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Results first posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Healthy Aging; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 2 arm, cross-sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate Intensity Aerobic Exercise (Experimental): 45-55% of heart rat reserve (HHR) Low range = ((Max HR from Visit 1) - Resting HR ) * 0.45 + Resting HR High range = ((Max HR from Visit 1) - Resting HR) * 0.55 + Resting HR
  Interventions: Behavioral: Aerobic Exercise
- High Intensity Aerobic Exercise (Experimental): 65-75% of heart rat reserve (HHR) Low range = ((Max HR from Visit 1) - Resting HR ) * 0.65 + Resting HR High range = ((Max HR from Visit 1) - Resting HR) * 0.75 + Resting HR
  Interventions: Behavioral: Aerobic Exercise

INTERVENTIONS:
Behavioral: Aerobic Exercise — Participants will exercise for 15 minutes based on heart rate range. The study team will employ a stationary bike to maintain control over workload

SUMMARY:
The overall goal is to characterize the acute exercise response as it relates to brain glucose metabolism in aging and Alzheimer's Disease (AD). The study team will also examine lactate metabolism, relationships with cognition, and the effect of exercise intensity.

DETAILED DESCRIPTION:
Aim 1: Compare the effects of acute, moderate intensity and acute, higher intensity exercise on cerebral glucose metabolism in nondemented (ND) elderly and AD subjects. ND (n=30) and AD (n=30) subjects will undergo a single bout of moderate intensity (45-55% HRR) or higher intensity (65-75% HRR) exercise to assess the effect of exercise intensity on acute change in brain glucose metabolism (rest to exercise). Investigators hypothesize that both moderate and high intensity exercise will elicit a drop in global brain glucose metabolism compared to quiet rest, but that the effect will be greater with higher intensity vs. moderate intensity exercise, and greater in ND subjects than in AD subjects.

Aim 2: Characterize the effect of both exercise intensities on acute biomarker response and cognition (memory and executive function) in ND and AD subjects. The acute biomarker response to exercise and the effect on cognition has not been examined in aged or AD cohorts. Investigators hypothesize that acute higher intensity exercise will elicit a greater blood lactate response (area under the curve, AUC) compared to acute moderate intensity exercise, and that this response will be greater in ND than in AD subjects. Investigators further hypothesize that lactate AUC will track negatively with change in cerebral glucose metabolism and cognitive performance. Although investigators will focus on lactate, they will also quantify additional exercise-related biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 and older
* Stable medication doses (>1month)
* Post-menopausal
* Diagnosis of either Nondemented (CDR 0) or Probable AD (CDR 0.5 or 1 only)

Exclusion Criteria:

* Inability to provide consent
* Diagnosis of insulin-dependent (Type 1) Diabetes Mellitus
* Recent ischemic heart disease (<2 years)
* Diagnosis of an clinically significant chronic disease including cardiovascular disease (CVD), other metabolic diseases (e.g., thyroid), cancer, human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome
* Excluded from or unable to complete an MRI scan
* Any Neurological disorders that have the potential to impair cognition or brain metabolism (e.g., Parkinson's disease, stroke defined as a clinical episode with neuroimaging evidence in an appropriate area to explain the symptoms).
* Clinically significant depressive symptoms that may impair cognition, abnormalities in B12, rapid plasma regain (RPR), or thyroid function that may impair cognition, use of psychoactive and investigational medications, and significant visual or auditory impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Green ZD, John CS, Kueck PJ, Blankenship AE, Kemna RE, Johnson CN, Yoksh LE, Best SR, Donald JS, Mahnken JD, Burns JM, Vidoni ED, Morris JK. Acute exercise alters brain glucose metabolism in aging and Alzheimer's disease. J Physiol. 2024 Sep 11:10.1113/JP286923. doi: 10.1113/JP286923. Online ahead of print. PMID 39258961
- [Background] Green ZD, John CS, Kueck PJ, Burns JM, Perry M, Donald J, Mahnken JD, Honea RA, Vidoni ED, Morris JK. Rationale and methods to characterize the acute exercise response in aging and Alzheimer's Disease: the AEROBIC pilot study. Contemp Clin Trials. 2021 Aug;107:106457. doi: 10.1016/j.cct.2021.106457. Epub 2021 May 27. PMID 34051350

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Moderate Intensity Aerobic Exercise | High Intensity Aerobic Exercise
Started | 29 | 31
Completed | 27 | 31
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — issue with PET image (1) | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Intensity Aerobic Exercise | High Intensity Aerobic Exercise | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 25 | 27 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.2 (7.3) | 74.2 (8.1) | 73.2 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 29
  Male | 16 | 15 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 2 | 6
  White | 24 | 29 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 31 | 60

OUTCOME MEASURES:

1. Primary Outcome: Fluorodeoxyglucose (FDG) Positron Emission Tomography (PET) Metabolism (Standard Uptake Value Ratio)
Description: FDG PET measures reflecting cerebral metabolism standardized to the uptake value of the cerebellum and standardized uptake value ratios (SUVR) calculated from native-space region of interest (ROI).
Time Frame: Resting Vs acute exercise bout: ~1 month
Measure: Mean (Standard Deviation); unit: SUVR
Arm/Group | Moderate Intensity Aerobic Exercise | High Intensity Aerobic Exercise
Number analyzed (Participants) | 27 | 31
SUVR | -0.0514 (0.03) | -0.0667 (0.03)

2. Secondary Outcome: Lactate Area Under the Curve
Description: Change in lactate AUC between the resting and exercise condition
Time Frame: Resting Vs acute exercise bout: ~1 month
Population: Individuals who completed both visits with blood draws available
Measure: Mean (Standard Deviation); unit: AUC change (mmol/L*min)
Arm/Group | Moderate Intensity Aerobic Exercise | High Intensity Aerobic Exercise
Number analyzed (Participants) | 28 | 31
AUC change (mmol/L*min) | 40.3 (27.5) | 97.0 (50.8)

3. Secondary Outcome: Brain-derived Neurotrophic Factor (BDNF) Change
Description: Pre/post change in circulating Brain Derived Neurotrophic Factor between the resting and exercise conditions
Time Frame: Resting Vs acute exercise bout: ~1 month
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Moderate Intensity Aerobic Exercise | High Intensity Aerobic Exercise
Number analyzed (Participants) | 28 | 31
pg/mL | 610.2 (1071.9) | 353.3 (239.8)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Moderate Intensity Aerobic Exercise | High Intensity Aerobic Exercise
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/31
Other Adverse Events (participants affected / at risk) | 2/29 | 2/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moderate Intensity Aerobic Exercise (N=29) | High Intensity Aerobic Exercise (N=31)
Abnormal ECG (Cardiac disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Covid diagnosis (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT04299308/Prot_SAP_000.pdf